CLINICAL TRIAL: NCT01097525
Title: Optical Quality, Threshold Target Identification, and Military Target Task Performance After Advanced Keratorefractive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fort Belvoir Community Hospital (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); US Army Night Vision and Electronic Sensors Directorate (Unknown)
Responsible Party: Principal Investigator, LTC Bruce Rivers, Director, Warfighter Refractive Eye Surgery Program and Research Center at FT Belvoir, Fort Belvoir Community Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20481
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Myopia; Myopic Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Wavefront guided (WFG) PRK (Active Comparator)
  Interventions: Procedure: WFG PRK
- WFG LASIK (Active Comparator)
  Interventions: Procedure: WFG LASIK
- Wavefront optimized (WFO) PRK (Active Comparator)
  Interventions: Procedure: WFO PRK
- WFO LASIK (Active Comparator)
  Interventions: Procedure: WFO LASIK

INTERVENTIONS:
Procedure: WFG PRK
  Arms: Wavefront guided (WFG) PRK
Procedure: WFG LASIK
  Arms: WFG LASIK
Procedure: WFO PRK
  Arms: Wavefront optimized (WFO) PRK
Procedure: WFO LASIK
  Arms: WFO LASIK

SUMMARY:
To determine the effect of two types of wavefront modalities (WFG vs. WFO) and two types of refractive surgery (PRK vs. LASIK) on visual and military task performance after laser refractive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy active adults with access to medical care at Walter Reed Health Care System.
2. Male or female at least 21 years old at the time of the pre-operative examination, and have signed an informed consent. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
3. Myopic spherical manifest refractive error from -1.00D up to -10.00D inclusive, with no more than 4.00D of manifest cylinder refractive error.
4. Inclusion based on pre-op Central Corneal Thickness (CCT) will be assessed according to Residual Stromal Bed Thickness
5. BSCVA of at least 20/20 in the study eye.
6. Soft contact lens users must have removed their lenses at least two weeks prior to baseline and follow-up measurements.
7. Hard contact lens users (PMMA or rigid gas permeable lenses) must have removed their lenses at least four weeks prior to baseline and follow-up measurements.
8. Refractive stability must be documented by previous refractions. Spherical and cylindrical portion of the manifest refraction must not have varied by more than 0.50 diopters over the previous 12 months.
9. Exhibits strong motivation for keeping the follow-up visits.
10. Available for evaluation at Walter Reed during the 1 year follow-up period
11. If selected, willing and available to undergo testing at Ft. Belvoir during the study period.
12. All service members must have a signed command authorization to receive government sponsored refractive surgery. The signed command authorization will be included in the original application.
13. Access to transportation to meet follow-up requirements.

Exclusion Criteria:

1. Residual, recurrent or active ocular diseases or congenital corneal abnormalities in either eye such as iritis, uveitis, keratoconjunctivitis sicca, herpetic keratitis, vernal conjunctivitis, lagophthalmos, corneal scarring, anterior basement membrane disease, recurrent erosions, glaucoma, previous steroid responder, occludable chamber angles, visually significant cataracts.
2. History of any previous eye surgery or trauma, including previous refractive surgery.
3. Dry eye as reflected by Schirmer's test, subjective complaints or symptoms of dry eye, findings during slit lamp exam that would be consistent with dry eye (e.g. superficial punctuate keratitis).
4. Corneal thickness insufficient to allow the residual remaining stromal bed to be no less than 300 microns in each eye. The residual stromal bed thickness will be determined by subtracting both the LASIK flap thickness and depth of the ablation from the total central corneal thickness measured by pachymetry.
5. Female subjects who are pregnant, breast-feeding or intend to become pregnant during the study. This is standard of care exclusion for refractive surgery at the Walter Reed Refractive Surgery Center because of the medications that are routinely given as part of the procedures. Standard of care analgesia consists of medications (e.g. narcotics) labeled as Pregnancy Category "C" by the FDA. Teratogenic effects are not known, however, physical dependence in the neonate may occur if the mother is given narcotics. Female subjects will be given a urine pregnancy test prior to participating in the study to rule out pregnancy.
6. Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin (Accutane), amiodarone hydrochloride (Cordarone) and/or sumatripin (Imitrex).
7. Significant corneal neovascularization.
8. Progressive myopia or keratoconus.
9. Medical condition(s), which, in the judgment of the investigator, may impair healing, including but not limited to: collagen vascular disease, autoimmune disease, immunodeficiency diseases, and ocular herpes zoster or simplex.
10. Patients with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course.
11. Any physical or mental impairment which would preclude participation in any of the examinations.
12. Inability to meet the mandated follow-up visit schedule for any reason such as duty hours, impending deployments, or PCS.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2010-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
visual outcomes | 12 months postoperatively
  Visual outcomes will be measured in terms of:
  * number of eyes achieving uncorrected visual acuity (UDVA) 20/20 or better.
  * number of eyes maintaining one Snellen line of corrected distance visual acuity (CDVA).
  * number of eyes within 0.50 diopter of manifest spherical equivalent.
objective image quality | 12 months postoperatively
  as measured by wavefront aberrometry
military task performance | 6 months postoperatively
  as measured by threshold target identification and night firing range
visual performance | 12 months postoperatively
  as measured by contrast sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Kraig S Bower, MD, Principal Investigator — The Wilmer Eye Institute, Johns Hopkins University
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia